CLINICAL TRIAL: NCT07246824
Title: Expanding Access to Safe Water in Nigeria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Princeton University (Other)
Responsible Party: Principal Investigator, Elisa Maria Maffioli, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00277959
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Chlorination
Keywords: Diarrhea; Health Systems
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Community Demonstrations and Redemption Points
  Interventions: Behavioral: Community Demonstrations; Behavioral: Redemption points
- Control (No Intervention): Neither community distributions will be conducted nor redemption points will be set-up during the study period

INTERVENTIONS:
Behavioral: Community Demonstrations — Facilitators will collaborate with local leaders, WASH officials and health facility staff in conducting community demonstrations introducing the chlorine product (WaterGuard+) to communities in the treatment group. Local leaders in the community will organize the meeting, while facilitators in the country will demonstrate how to use the product, what the correct dosage is, and explain the importance of water treatment. They will also show how village water is contaminated with Ecoli. These meetings will be targeted at eligible women (pregnant women and women with children under the age of 5), however all members of the community will be invited to attend. At the meeting, each attendee will be given one bottle of WaterGuard+, which is enough to treat drinking water for a household of 5 members for about a month, and 1,000 naira. Water Guard + is a 180g bottle of sodium dichloroisocyanurate (NaDCC) in granulated / powder form, produced and distributed by the Society for Family Health.
  Arms: Treatment
Behavioral: Redemption points — Study staff will set up at least one chlorine redemption point for each community. The location of the redemption point will be determined in consultation with the local community during Community Demonstrations. The redemption points could be health facilities, local shops/dispensaries/kiosks, local pharmacies, house of the village leader, CHW, or health staff or other suitable sites. Households will be able to visit the location and redeem a month's supply of a chlorine product. Distributors will use a redemption log to keep track of when participants redeem the chlorine product.
  Arms: Treatment

SUMMARY:
Access to safe water remains a pressing public health challenge in Nigeria, where 67% of the population lacks safely managed drinking water and waterborne diseases cause an estimated 70,000 child deaths annually. Building on evidence that point-of-use chlorination is highly cost-effective in reducing diarrheal disease, this study evaluates a scalable, community-based chlorine distribution model through a cluster-randomized controlled trial (RCT) in Kano State. Thirty communities across four Local Government Areas will be randomly assigned to one of three groups: (i) 20 treatment communities receiving community demonstrations and local chlorine redemption points, (ii) 10 control communities where no intervention will be conducted. After 3 months, 5 control communities will receive an individual-level sensitization and a voucher program and 5 will remain pure control communities. The RCT aims to estimate the causal impact of the community-based intervention on household chlorination rates, water quality (E. coli contamination), and knowledge of safe water practices over six months. By rigorously testing a community-led water treatment model, this study contributes new evidence on sustainable and cost-effective approaches to expand safe water access in low-resource settings. The results will inform national and regional strategies for scaling point-of-use chlorination across sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers and women with children under 5 children

Exclusion Criteria:

* Men, women with no children under 5 years old

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 700 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Treat drinking water with chlorine (tested in water sample) | Measured up to 6 months of follow-up
  Proportion of water samples with detectable chlorine in stored drinking water

SECONDARY OUTCOMES:
Treat drinking water with chlorine (self-reported) | Measured up to 6 months of follow-up
  Proportion of women who reported using chlorine in the previous two days
Presence of E.coli | Measured up to 6 months of follow-up
  Proportion of water samples with detectable E.coli
Level of E.coli | Measured up to 6 months of follow-up
  Level of E-coli (in log10 MPN/100ml) in water samples
Unsafe risk of Coliform | Measured up to 6 months of follow-up
  Proportion of water samples with unsafe coliform ( >100 colony forming units per 100mL)
Heard about chlorine | Measured up to 6 months of follow-up
  Proportion of women who ever heard about chlorine
Ever used chlorine | Measured up to 6 months of follow-up
  Proportion of women who ever used chlorine
Last used chlorine | Measured up to 6 months of follow-up
  Proportion of women who used chlorine yesterday or the day before

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Maria Maffioli, PhD, Principal Investigator — University of Michigan; Pascaline Dupas, Principal Investigator — Princeton University; Ana Radu, Principal Investigator — Princeton University
Locations (1):
- Kura, Dawakin Kudu, Kiru, and Rano LGAs, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: No